CLINICAL TRIAL: NCT01909063
Title: A Randomized Controlled Trial Testing the Effect of a Multi-nutrient Fortified Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Michael F. Holick, Principal Investigator, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Multinutrient Fortified Juice
Record Dates: First submitted 2012-06-25; First posted 2013-07-26 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Vitamin D Deficiency; Hypovitaminosis A; Vitamin E Deficiency
MeSH Terms: conditions — Vitamin D Deficiency; Avitaminosis; Vitamin E Deficiency | interventions — Vitamin D; Vitamin E; Vitamin A; Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): 200 IU vitamin D and 700 mg of calcium per day in 2 glasses of juice per day for 2 weeks
  Interventions: Dietary Supplement: Vitamin D
- Arm B (Experimental): 200 IU vitamin D, 12 IU vitamin E, 2000 IU vitamin A as beta carotene, and 700 mg of calcium per day in 2 glasses of juice
  Vitamin D, Vitamin E, and Vitamin A
  Interventions: Dietary Supplement: Vitamin D, Vitamin E, and Vitamin A
- Arm C (Placebo Comparator): Control, 700 mg of calcium per day in 2 glasses of juice
  Control, 700 mg Calcium
  Interventions: Dietary Supplement: Control, 700 mg Calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D — Fortification of orange juice with 200 IU vitamin D to be drunk twice per day for 12 weeks
  Arms: Arm A
Dietary Supplement: Vitamin D, Vitamin E, and Vitamin A — Fortification of orange juice with Vitamin D, Vitamin E, and Vitamin A to be drunk twice per day for 12 weeks
  Arms: Arm B
Dietary Supplement: Control, 700 mg Calcium — Orange juice with 700 mg calcium to be drunk twice per day for 12 weeks
  Arms: Arm C

SUMMARY:
The goal of this investigator-initiated study is to determine whether the fortification of orange juice with vitamin D, vitamin A, and vitamin E will enhance the vitamin D, vitamin A, and vitamin E status children ages 6-10 that are seen at the Division of Pediatrics at Boston University Medical Center. Circulating concentrations of 25-hydroxyvitamin D [25(OH)D], vitamin A, and vitamin E before, will be measured at mid-intervention (week 6), and after a period of twelve weeks. This study plans to recruit 180 male and female subjects between the ages of 6 and 10. An informed consent will be explained and discussed with the subjects and their parents/guardians willing to participate in the study. The study will be twelve weeks. Blood will be drawn during the initial visit, mid-intervention (week 6), and week 12. Dietary intake will be assessed at baseline and at the conclusion of the 12-week intervention using a 3-day food record. The subjects will be randomized in a double-blinded manner via an electronically shuffled listed. Subjects will be randomized to receive one of three beverages: (1) calcium plus vitamin D fortified orange juice (intervention A), (2) calcium plus vitamins D, A, and E fortified orange juice (intervention B) or (3) calcium-only fortified orange juice (controls). Subjects in all groups will drink two 8-oz. glasses of juice at least six hours apart (morning and afternoon) per day for a period of 12 weeks. Subjects randomized to intervention A will receive 200 IU vitamin D and 700 mg of calcium per day in 2 glasses of juice, intervention B will receive 200 IU vitamin D, 12 IU vitamin E, 2000 IU vitamin A as beta carotene, and 700 mg of calcium per day in 2 glasses of juice, while controls will receive 700 mg of calcium per day in 2 glasses of juice. A blood sample will be obtained before the subjects begin drinking the orange juice and at week 12 to determine levels of 25(OH)D which is a measure of vitamin D status. Blood will also be used for determining osteocalcin, parathyroid hormone (PTH), alkaline phosphatase, phosphorus, calcium, C-telopeptide (CTX), albumin, vitamin A, and vitamin E. A blood sample will also be obtained at week 6 for 25(OH)D and PTH.

DETAILED DESCRIPTION:
This is an investigator-initiated double-blinded study in which one hundred and eighty male and female subjects ages 6 to 10 will be recruited from the Division of Pediatrics at Boston University Medical Center. Potential volunteers will undergo a screening process to ensure that inclusion and exclusion criteria are met. A general medical history will be taken before the study starts. A baseline biochemical profile (blood) including calcium, phosphorus, osteocalcin, alkaline phosphatase, C-telopeptide (CTX), 25(OH)D, PTH, albumin, vitamin A, and vitamin E will be determined after the study is completed. The amount of blood estimated to be drawn on the first visit is 27 ml. Dietary intake will be assessed from 3 day food records via NDS-Minnesota Database by Dr. Christine Economos, Friedman School of Nutrition Science and Policy at Tufts University. Once the subject has met the inclusion criteria, he/she will receive two gallons of orange juice via a delivery service to their home. He/she will be instructed to drink two 8 oz. glasses of orange juice a day and record each glass of juice that was drunk; stickers and calendars will be provided. A delivery service will be used to deliver juice to parents/caregiver biweekly. Signature and log sheets of deliveries will be maintained. A glass that has a mark designating eight ounces will be provided to the subject so that the amount of orange juice that is drunk is measured. Sixty subjects will receive intervention A, sixty subjects will receive intervention B, and sixty subjects will receive intention C. Subjects randomized to intervention A will receive juice that contains 200 IU of vitamin D and 700 mg of calcium per day. Subjects randomized to intervention B will receive 200 IU vitamin D, 12 IU vitamin E, 2000 IU vitamin A as beta-carotene, and 700 mg of calcium per day. Subjects randomized to intervention C will receive 700 mg calcium per day. A venous blood sample of 27 ml [two red top tubes (10ccs each) and one purple top tube (7ccs)] will be obtained at the initial and final visits. 25(OH)D, PTH, calcium, phosphorus, osteocalcin, C-telopeptide(CTX), alkaline phosphatase, albumin, vitamin A, and vitamin E will be measured from the blood samples. During the mid-intervention blood draw (week 6) 10mL of blood will be drawn and 25(OH)D and PTH will be measured. The study will consist of 12 weeks of drinking two eight-ounce glasses of orange juice a day (one in the am and one in the pm).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female children of all races with ages between 6 and 10

Exclusion Criteria:

1. History of rickets
2. History of intestinal malabsorption (i.e. Cystic Fibrosis, Fat Malabsorption Syndrome, Crohn's Disease)
3. History of severe medical illness, including renal failure (decrease 2/3 kidney function)
4. Allergies to orange juice
5. Any medical conditions in which it is not advisable to receive two 8 oz. glasses of orange juice per day
6. History of Diabetes
7. Currently taking, or having taken less than one month prior to start of study, a prescription vitamin D
8. Unwilling to consent/assent to this trial

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Improve Vitamin A, Vitamin E, and Vitamin D Status in Children | 12 weeks
  The primary outcome of this study is to determine if fortification of orange juice with vitamin D, vitamin A, and vitamin E will enhance the vitamin D, vitamin A, and vitamin E status children ages 6-10 that are seen at the Division of Pediatrics at Boston University Medical Center.

CONTACTS AND LOCATIONS:
Overall Officials: Micahel F Holick, PhD, MD, Principal Investigator — BUMC
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States